CLINICAL TRIAL: NCT05888766
Title: How to Predict Response to Acute Treatment of Migraine With Rimegepant 75 mg: a Biochemical and Neurophysiological Study.
Brief Title: Predict the Response to Acute Treatment of Migraine With Rimegepant 75 mg
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gabriele Sebastianelli, Dr., University of Roma La Sapienza
Other Study IDs: S-LT-000002620231
Record Dates: First submitted 2023-05-07; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Migraine Disorders
Keywords: migraine biomarkers; neurophysiology; CGRP; salivary CGRP; habituation; sensitization; Rimegepant
MeSH Terms: conditions — Migraine Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Salivary samples where CGRP concentration will be quantified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Episodic migraine patients: 20 patients with episodic migraine (<15 attacks/month) will be recruited from a specialized headache Clinic (headache clinic of the Sapienza University of Rome, Latina).
  Interventions: Drug: Rimegepant 75 milligrams

INTERVENTIONS:
Drug: Rimegepant 75 milligrams — At the screening visit patients with episodic migraine, which will be prescribed Rimegepant 75 mg as abortive treatment, will be asked to participate in the study.

SUMMARY:
Tools to predict which patients could better respond to abortive CGRP target therapy are still lacking. We propose to investigate if biochemical (salivary CGRP) and neurophysiological (evoked potentials) biomarkers can recognize patients with the best chances of responding to Rimegepant 75 mg as an acute treatment of migraine.

DETAILED DESCRIPTION:
Background: The understanding of the central role of CGRP in migraine pathophysiology led to the development of new target therapies against this molecule pathway, including Rimegepant. Despite the central role of the CGRP pathway in migraine, it was recently discovered that some migraine attacks are non CGRP-dependent. Tools to predict which patients could better respond to abortive CGRP target therapy are still lacking.

Objective: We propose to investigate if biochemical (salivary CGRP) and neurophysiological (evoked potentials) biomarkers can recognize patients with the best chances of responding to Rimegepant 75 mg as an acute treatment of migraine.

Design of the study and methods: This will be a prospective observational study. The study will be subdivided into four phases: screening visit (T0), salivary collection, observational phase, follow-up visit (T1). At the screening visit (T0) patients with episodic migraine (20 patients), which will be prescribed Rimegepant 75 mg as abortive treatment, will be asked to participate in the study. During the salivary collection phase, patients will be instructed to collect daily saliva samples for a minimum of 7 days and a maximum of 14 days to include a minimum of 1 migraine attack. During the observational phase (1-month duration) patients will take Rimegepant 75 mg for abortive treatment of migraine attacks and, they will be instructed to take extra saliva samples (headache onset, after 2h and 8h) at each migraine attack. Neurophysiological procedures (somatosensory evoked potentials and nociceptive blink reflex) will be recorded at baseline (T0) and after 1 month (follow-up visit, T1) of administration of Rimegepant 75 mg as an abortive migraine treatment. We chose somatosensory evoked potentials (SSEPs) to assess the integrity of the non-pain-related somatosensory lemniscal system and to study habituation phenomena, and nociceptive blink reflex (nBR) to investigate the activity of the caudal trigeminal nucleus. CGRP salivary levels will be quantified with ELISA kit.

Specific aim: We aim to predict Rimegepant (used as abortive therapy) response from baseline CGRP salivary levels and neurophysiological parameters (habituation and sensitization from somatosensory evoked potentials and nociceptive blink reflex). Mixing and comparing these two approaches could help to find a combination of biomarkers able to predict the treatment success. We hypothesize that patients with marked habituation deficit, less sensitization, and more elevated CGRP salivary levels during the attack will be the patients who will respond the most to Rimegepant 75 mg as abortive migraine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Episodic migraine
* Prescription of Rimegepant 75 mg as abortive treatment for migraine
* headache occurring on < 15 days/four weeks;
* No other primary/secondary headache disorder;
* No contraindication for Rimegepant 75 mg;
* No previous exposure to any anti-CGRP drugs;
* No prophylactic migraine treatment ongoing or in the past 3 months before participation in the study

Exclusion Criteria:

* headache occurring >15 days/four weeks
* Contraindication for Rimegepant 75 mg
* Previous exposure to anti-CGRP drugs;
* Prophylactic migraine treatment ongoing or in the past 3 months before participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients with episodic migraine recruited from a specialized headache Clinic (headache clinic of the Sapienza University of Rome, Polo-Pontino ICOT, Latina).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Salivary CGRP levels during attacks | from enrollment to one month after the start of therapy
  In order to identify a biomarker that predicts the Rimegepant's response
Relationship between Rimegepant's response and salivary CGRP levels | from enrollment to one month after the start of therapy
  Differences between responders and not responders to Rimegepant and salivary CGRP levels (pg/ml).
Relationship between Rimegepant's response and habituation at baseline | from enrollment to one month after the start of therapy
  Differences between responders and not responders to Rimegepant and habituation (microvolt) at baseline.
Relationship between Rimegepant's response and sensitization at baseline | from enrollment to one month after the start of therapy
  Differences between responders and not responders to Rimegepant and sensitization (microvolt) at baseline.

SECONDARY OUTCOMES:
Effects of Rimegepant 75 mg on habituation after 1 month of therapy | one month after the start of therapy
  Comparison between habituation (microvolt) at baseline and habituation (microvolt) after one month of abortive therapy with Rimegepant 75 mg
Changes from Baseline in the sensitization after 1 month of therapy | one month after the start of therapy
  Comparison between sensitization (microvolt) at baseline and sensitization (microvolt) after one month of abortive therapy with Rimegepant 75 mg
Changes from Baseline in the pain threshold after 1 month of therapy | one month after the start of therapy
  Comparison between pain threshold (mA) at baseline and pain threshold (mA) after one month of abortive therapy with Rimegepant 75 mg
Changes from Baseline in the sensory detection threshold after 1 month of therapy | one month after the start of therapy
  Comparison between sensory detection threshold (mA) at baseline and sensory detection threshold (mA) after one month of abortive therapy with Rimegepant 75 mg

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Sebastianelli, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome Polo Pontino - ICOT, Latina, Italy / Latina, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Croop R, Goadsby PJ, Stock DA, Conway CM, Forshaw M, Stock EG, Coric V, Lipton RB. Efficacy, safety, and tolerability of rimegepant orally disintegrating tablet for the acute treatment of migraine: a randomised, phase 3, double-blind, placebo-controlled trial. Lancet. 2019 Aug 31;394(10200):737-745. doi: 10.1016/S0140-6736(19)31606-X. Epub 2019 Jul 13. PMID 31311674
- [Result] Lipton RB, Croop R, Stock EG, Stock DA, Morris BA, Frost M, Dubowchik GM, Conway CM, Coric V, Goadsby PJ. Rimegepant, an Oral Calcitonin Gene-Related Peptide Receptor Antagonist, for Migraine. N Engl J Med. 2019 Jul 11;381(2):142-149. doi: 10.1056/NEJMoa1811090. PMID 31291516
- [Result] Alpuente A, Gallardo VJ, Asskour L, Caronna E, Torres-Ferrus M, Pozo-Rosich P. Salivary CGRP can monitor the different migraine phases: CGRP (in)dependent attacks. Cephalalgia. 2022 Mar;42(3):186-196. doi: 10.1177/03331024211040467. Epub 2021 Oct 4. PMID 34601944
- [Result] Ashina M, Terwindt GM, Al-Karagholi MA, de Boer I, Lee MJ, Hay DL, Schulte LH, Hadjikhani N, Sinclair AJ, Ashina H, Schwedt TJ, Goadsby PJ. Migraine: disease characterisation, biomarkers, and precision medicine. Lancet. 2021 Apr 17;397(10283):1496-1504. doi: 10.1016/S0140-6736(20)32162-0. Epub 2021 Mar 25. PMID 33773610
- [Result] Alpuente A, Gallardo VJ, Asskour L, Caronna E, Torres-Ferrus M, Pozo-Rosich P. Salivary CGRP and Erenumab Treatment Response: Towards Precision Medicine in Migraine. Ann Neurol. 2022 Nov;92(5):846-859. doi: 10.1002/ana.26472. Epub 2022 Aug 24. PMID 36054144
- [Result] Messlinger K, Vogler B, Kuhn A, Sertel-Nakajima J, Frank F, Broessner G. CGRP measurements in human plasma - a methodological study. Cephalalgia. 2021 Nov;41(13):1359-1373. doi: 10.1177/03331024211024161. Epub 2021 Jul 16. PMID 34266288
- [Result] Casillo F, Sebastianelli G, Di Renzo A, Cioffi E, Parisi V, Di Lorenzo C, Serrao M, Coppola G. The monoclonal CGRP-receptor blocking antibody erenumab has different effects on brainstem and cortical sensory-evoked responses. Cephalalgia. 2022 Oct;42(11-12):1236-1245. doi: 10.1177/03331024221103811. Epub 2022 May 30. PMID 35637558
- [Result] Sebastianelli G, Casillo F, Di Renzo A, Abagnale C, Cioffi E, Parisi V, Di Lorenzo C, Serrao M, Pierelli F, Schoenen J, Coppola G. Effects of Botulinum Toxin Type A on the Nociceptive and Lemniscal Somatosensory Systems in Chronic Migraine: An Electrophysiological Study. Toxins (Basel). 2023 Jan 14;15(1):76. doi: 10.3390/toxins15010076. PMID 36668895
- [Result] Coppola G, Di Lorenzo C, Schoenen J, Pierelli F. Habituation and sensitization in primary headaches. J Headache Pain. 2013 Jul 30;14(1):65. doi: 10.1186/1129-2377-14-65. PMID 23899115